CLINICAL TRIAL: NCT01589354
Title: Effectiveness of Interscalene Brachial Plexus Block and Intra-articular Injection of Ropivacaine for Post-operative Analgesia in Arthroscopic Shoulder Stabilization Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Grampian (Other Government)
Responsible Party: Principal Investigator, Amr M Mahdy, Dr, NHS Grampian
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10/S0801/74
Record Dates: First submitted 2012-04-29; First posted 2012-05-01 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Postoperative Analgesia
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interscalene brachial plexus block (Experimental)
  Interventions: Procedure: Interscalene brachial plexus block; Device: Ultrasound guided technique; Drug: Ropivacaine
- Intra-articular injection (Experimental)
  Interventions: Procedure: Intra-articular Ropivacaine injection; Drug: Ropivacaine

INTERVENTIONS:
Procedure: Interscalene brachial plexus block — An interscalene block will be performed pre-operatively using ultrasound guidance and the peripheral nerve stimulator (with the patient awake) using 20 ml of 0.375% Ropivacaine.
  Arms: Interscalene brachial plexus block
Procedure: Intra-articular Ropivacaine injection — The procedure will be done by the surgeon at the end of the operation, with an intra-articular injection of 20 ml 0.75% Ropivacaine through the arthroscopic cannula after closure of the anterior wound
  Arms: Intra-articular injection
Device: Ultrasound guided technique — The block will be performed under U/S guidance
  Arms: Interscalene brachial plexus block
Drug: Ropivacaine — 20ml of 0.375% Ropivacaine
  Arms: Interscalene brachial plexus block
Drug: Ropivacaine — 20ml of 0.75% Ropivacaine injected by the surgeon at the end of the procedure
  Arms: Intra-articular injection

SUMMARY:
This study evaluates two anaesthetic techniques namely interscalene brachial plexus block and intra-articular local anaesthetic injection. Both techniques are currently used for providing postoperative pain relief following arthroscopic shoulder stabilisation operation. It will be a randomised controlled trial involving 30 patients in two groups.

ELIGIBILITY:
Inclusion Criteria:

• All adult patients above the age of 18 years undergoing arthroscopic shoulder stabilisation operation

Exclusion Criteria:

* Patients not meeting inclusion criteria
* Patients unable to give informed consent
* Patient refusal to participate in the study
* Contraindications to Interscalene block
* Allergy to local anaesthetics
* Peripheral neuropathy from any cause
* Patients on opiates for chronic pain
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Mean pain score over the first 24 hours following arthroscopic shoulder stabilisation operation | 24 months

SECONDARY OUTCOMES:
Post-operative analgesic requirements in the first 24 hours after surgery | 24 months
Patient assessment of quality of analgesia and identifying any complications as a result of the two anaesthetic procedures | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Amr M Mahdy, MD, Principal Investigator — NHS Grampian